CLINICAL TRIAL: NCT06903338
Title: A Phase 3 Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Tobevibart + Elebsiran Combination Therapy in Participants With Chronic HDV Infection (ECLIPSE 1)
Brief Title: A Study to Evaluate Tobevibart + Elebsiran in Chronic HDV Infection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-CHDV-V203
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Viral Hepatitis
Keywords: HDV; Hepatitis D Virus; Hepatitis; Chronic Hepatitis D Virus; Hepatitis D; Hepatitis D, Chronic; Hepatitis Delta Virus
MeSH Terms: conditions — Hepatitis; Hepatitis D; Hepatitis D, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Tobevibart + Elebsiran) (Experimental): Participants will receive treatment with tobevibart + elebsiran for 240 weeks.
  Interventions: Drug: Tobevibart; Drug: Elebsiran
- Arm 2 (Tobevibart + Elebsiran) (Experimental): Participants will receive tobevibart + elebsiran after an observational period for 240 weeks.
  Interventions: Drug: Tobevibart; Drug: Elebsiran

INTERVENTIONS:
Drug: Tobevibart — Tobevibart administered by subcutaneous injection
  Other Names: VIR-3434
Drug: Elebsiran — Elebsiran administered by subcutaneous injection
  Other Names: VIR-2218

SUMMARY:
This is a multicenter, open label, randomized Phase 3 clinical study to evaluate the efficacy and safety of the combination of tobevibart + elebsiran for the treatment of chronic hepatitis delta in comparison to delayed treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 18 to 70 years at screening
2. Chronic HDV infection for >/= 6 months
3. On NRTI therapy against HBV for at least 12 weeks prior to day 1 or have HBV DNA < 20 IU/ml at screening, currently on locally approved NRTI therapy
4. Serum ALT > ULN and < 5x ULN
5. Non-cirrhotic or Compensated Cirrhotic Liver Disease at screening

Exclusion Criteria:

1. Any clinically significant chronic or acute medical or psychiatric condition that makes the participant unsuitable for participation.
2. History of significant liver disease from non-HBV or non-HDV etiology
3. History of allergic reactions, hypersensitivity, or intolerance to study drug, its metabolites, or excipients.
4. History of anaphylaxis
5. History of immune complex disease
6. History of autoimmune disorder
7. History or evidence of alcohol or drug abuse within 6 months before screening or a positive drug screen at screening unless it can be explained by a prescribed medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
HDV RNA < Lower Limit of Quantification (LLOQ), Target Not Detected (TND) and alanine aminotransferase (ALT) normalization (ALT </= Upper Limit of Normal [ULN]) at Week 48 for Arm 1 vs at Week 12 for Arm 2 | Up to 48 weeks
Incidence of Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) through Week 12 | Up to 12 weeks

SECONDARY OUTCOMES:
HDV RNA < LLOQ, TND at Week 48 for Arm 1 vs Week 12 for Arm 2 | Up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- United States (11):
  - Investigative Site, Chandler, Arizona
  - Investigative Site, Los Angeles, California
  - Investigative Site, Redwood City, California
  - Investigative Site, San Francisco, California
  - Investigative Site, DeLand, Florida
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Hillsborough, New Jersey
  - Investigative Site, New York, New York
  - Investigative Site, Murray, Utah
  - Investigative Site, Seattle, Washington
- Canada (6):
  - Investigative Site, Calgary, Alberta
  - Investigative Site, Montreal, Quebec
  - Investigative Site, Montreal
  - Investigative Site, Ottawa
  - Investigative Site, Québec
  - Investigative Site, Vancouver
- Investigative Site, Tbilisi, Georgia
- Germany (3):
  - Investigative Site, Frankfurt
  - Investigative Site, Hanover
  - Investigative Site, Heidelberg
- Investigative Site, Chisinau, Moldova
- Investigative Site, Auckland, New Zealand
- Pakistan (3):
  - Investigative Site, Karachi
  - Investigative Site, Lahore
  - Investigative Site, Rawalpindi
- Investigative Site, Bucharest, Romania
- Investigative Site, Kyiv, Ukraine
- United Kingdom (3):
  - Investigative Site, London
  - Investigative Site, Manchester
  - Investigative Site, Nottingham